CLINICAL TRIAL: NCT03129633
Title: Raices: A Promotores Network to Improve the Health Behaviors and Health Outcomes of Latino Immigrants Living in an Emerging Latino Community
Brief Title: Raices: A Promotores Network to Improve Latino Immigrant Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sharon Ross, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PRO17020357
Record Dates: First submitted 2017-04-07; First posted 2017-04-26 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promotores Network (Experimental): Promotores will engage participants using the materials A Page of My Life and the Success Plan. Promotores will ask participants to rank their satisfaction with each of the domains included in the A Page of My Life and ask them what domain they want to change. Using non-directive questions, promotores will guide the participant to draft a plan for success. The promotor/a will follow up with participants within a week of enrollment and at least monthly via phone/text during six months. During the intervention period, promotores will meet with participants (child and parent together, if applicable) at least three times in-person during which they will deliver the short (15-minutes) educational components of the intervention.
  Interventions: Other: Intervention group
- Wait-list Control (No Intervention): The community liaison will deliver a short (15-minute) educational session on the benefits of a healthy lifestyle and preventive use of health care, and give participants a pamphlet with relevant local health care and social service resources.

INTERVENTIONS:
Other: Intervention group — One-on-one contact with a promotor(a) over the 6 month intervention.
  Arms: Promotores Network

SUMMARY:
This study examines the effectiveness of a community health worker (promotores) network in improving access to care, social support, physical activity and nutrition in Latino immigrants living in an emerging Latino community.

DETAILED DESCRIPTION:
This proposal examines the potential of a community health worker (CHW) network to improve health behaviors and health outcomes of Latino immigrants living in an Emerging Latino Community (ELC; areas with low (<5%), yet growing concentrations of Latinos).CHWs (promotores in Spanish) are trained individuals from the community who establish interpersonal connections to reach and serve Latinos and address health disparities.

This proposal builds on two pilot studies conducted by the investigative team: (1) a community-based intervention delivered by promotores to increase social support and health care access in immigrant men, and (2) a home-based intervention delivered by promotoras to improve nutrition and physical activity in Latino preschool children and their families.

Little is known about the potential usefulness of a promotores network in improving both health care access and engagement in physical activity and healthy eating, compared with standard informational approaches, among Latino immigrants from an ELC. The proposed research will address the following specific aims:

(Sp. Aim 1) Develop and implement a structured, promotor/a-mediated intervention to increase access to care, social support, and engagement in health-promoting behaviors; (Sp. Aim 2) Examine the feasibility of a structured, promotor/a-mediated approach to peer support, with a participant-guided goal-setting component; and (Sp. Aim 3) Assess the effectiveness of a promotores network on increasing access to care, social support, and engagement in health-promoting behaviors compared with a waitlist-control group. Partnering with a federally-qualified health center and a social service organization, the investigators propose to employ a quasi-experimental design to assess the effect of a promotores network on outcomes measured at 6 months after enrollment, compared with a wait-list control.

The research team will hire and train 16 promotores and 8 community liaisons to recruit, assess, and deliver the intervention (promotores only). Participants will include adults and children (≥ 11 years) drawn from Allegheny County, Pennsylvania (an ELC). Promotores and RIs will recruit n=200 intervention and n=200 control participants using similar protocols from our pilot studies (e.g., word-of-mouth, flyers). The 6 month intervention will include using motivational interviewing techniques and intervention tools adapted from our previous work, to assist promotores in eliciting the participants' most important needs drawn from 8 life domains (e.g., health care, exercise/recreation, social life).

Promotores will guide the participant to set goals and follow-up over the 6 month intervention period (in-person and via phone) to measure progress, address barriers, and deliver short educational (health promotion) sessions.

Process evaluation includes a comprehensive set of questions to assess fidelity, dose, reach, recruitment and contextual factors using multiple data sources. Primary outcomes include access to care (preventive and usual source of care), social support, physical activity, and dietary intake. Expected outcomes include: (1) gain valuable information surrounding feasibility and effectiveness of proposed intervention protocol, (2) contribute to improving access to care and increasing health-promoting behaviors in Latinos living in an ELC, and (3) contribute to reducing health disparities in Latino individuals and families. The objectives of this project are in line with both the CMS mission of promoting better care, healthier people, and smarter spending for beneficiaries, and the Healthy People 2020 goals of eliminating disparities. This proposal carries high public health significance because it targets Latino health disparities through primary prevention and a structured approach to peer support, as well as maximizes the potential of both men and women promotores to assist participants living in an ELC

ELIGIBILITY:
Inclusion Criteria:

1. are between 2 -18 years of age (children) or ≥ 18 years of age (adult),
2. self-identify as Hispanic/Latino,
3. speak English/Spanish, and
4. live in Allegheny County, Pennsylvania.

Exclusion Criteria:

1. non-Hispanic/Latino,
2. primary language other than Spanish or English, or
3. cognitive limitation to complete surveys or interviews.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in number of participants who have access to care | 6 months
  # of participants having any health insurance, usual source of care, visit to Dr. or visit to dentist.
Change in Social Support | 6 months
  12-item scale
Change in Physical Activity levels | 6 months
  Min/day of self-reported moderate-to-vigorous physical activity:
Change in Dietary Behaviors | 6 months
  Usual Dietary intake

SECONDARY OUTCOMES:
Change in BMI | 6 months
  calculated using standard equation (kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon E Ross, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States